CLINICAL TRIAL: NCT01911650
Title: A Pilot Study Correlating Novel Ultrasound Elastography Techniques to Standard Clinical Outcomes in the Treatment of Achilles Tendinopathy With Platelet-Rich Plasma Therapy
Brief Title: A Pilot Study: Treatment of Achilles Tendinopathy With Platelet-Rich Plasma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-0908
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Achilles Tendinitis
Keywords: Achilles; tendinopathy
MeSH Terms: conditions — Tendinopathy | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Platlet Rich Plasma (Experimental): This subject arm will receive one injection of autologous platelet rich plasma for the treatment of Achilles tendinopathy. In addition, they will be asked to undergo a palpatory exam of the Achilles tendon; complete Quality of Life Questionnaires at three different time points; and complete a 30 minute ultrasound imaging exam of the Achilles tendon.
  Interventions: Other: Autologous Platelet Rich Plasma; Other: Ultrasound Imaging; Other: Quality of Life Questionnaires
- Waitlist (Other): Subjects in this arm will have already received standard of care interventions for Achilles tendinopathy with unsatisfactory outcomes. For this research they will be asked to undergo a palpatory exam of the Achilles tendon; complete Quality of Life Questionnaires at three different time points; and complete a 30 minute ultrasound imaging exam of the Achilles tendon.
  Interventions: Other: Ultrasound Imaging; Other: Quality of Life Questionnaires

INTERVENTIONS:
Other: Autologous Platelet Rich Plasma — This procedure will include a single collection of 35 mL of peripheral blood. A two-stage spinning protocol will be used: the 1st separates red blood cells from platelets, and the 2nd concentrates the platelets to yield approximately 4 mL of concentrated autologous platelet. This layer of platelet rich plasma will be placed in the syringe by the centrifuge machine.
  Arms: Autologous Platlet Rich Plasma
Other: Ultrasound Imaging — A conventional ultrasound in addition to AE and shear wave imaging (SWI) will be administered.
Other: Quality of Life Questionnaires — This questionnaire is a self-report of pain and function associated with the Achilles tendon.
  Other Names: Victorian Institute of Sports Assessment - Achilles (VISA-A)

SUMMARY:
The overall goal of this proposal is to correlate ultrasound elastography technique with more standard clinically based outcome measures within the setting of a small sample sized group of patients affected by moderate-to- severe, chronic (>6months) midsubstance Achilles tendinopathy (AT).

DETAILED DESCRIPTION:
The main goal for this pilot level study is to correlate ultrasound elastography technique with more standard clinically based outcome measures within the setting of a small sample sized group of patients affected by moderate-to- severe, chronic (> 6 months) midsubstance Achilles tendinopathy (AT). Investigators will conduct a 24-week, 2-arm randomized controlled pilot study to determine whether novel elastography techniques (AE) and shear wave imaging (SWI), a new quantitative method of ultrasound (US) imaging, correlate with valid clinical outcome measures (VISA-A and conventional US). Methods will be based on recently published clinical trials of autologous blood injections for treating AT and will incorporate novel US outcome measures of Achilles tendon appearance and stiffness, i.e. elasticity. The results of this multi-disciplinary pilot study will be used to help plan a separate larger scaled study to evaluate the effects of platelet-rich plasma (PRP) therapy for Achilles tendinopathy in which elastography will be included as a potential outcome measure and also correlated with standard clinical outcome surveys.

Pain and function will be evaluated by self-report using a validated clinical outcome questionnaire (VISA-A). Disease modification will be assessed by novel US-based AE and SWI methods for stiffness changes (biomechanical) and correlated with morphologic changes using conventional US. A larger study that will evaluate the effects of PRP in healing AT, while correlating with elastography assessment, will include a sham injection arm.

Intervention Subjects assigned to the PRP group will then receive the PRP injection under ultrasound guidance. The injection will take about 15 minutes.

Each subject will undergo a palpatory and ultrasound Achilles tendon exam. Tender areas associated with the Achilles tendon will be identified. Physical exam will be followed by Achilles tendon ultrasound which will serve as visual guidance for injection.

At the injection session, the research nurse will perform a single standard antecubital blood draw (35 mL). The PRP will be obtained from this sample using a two-stage spinning technique: the 1st separates red blood cells from platelets, and the 2nd concentrates the platelets to yield approximately 4 mL of concentrated autologous platelet. This layer of platelet rich plasma will be placed in the syringe by the centrifuge machine.

Platelet counts of subjects' whole blood and PRP processed blood will be analyzed. Platelet counts in whole blood vary by individual. The optimal quantity of platelets and growth factors required for tissue healing is not known, but a clinically effective concentration has been described as being greater than 4 times baseline autologous whole blood platelet concentrations. Therefore, platelet concentration yield may have important implications in clinical outcome correlation. In order to validate consistent platelet concentration yields across subjects, investigators will sample 1 mL of whole blood (approximately one lab Vacutainer) and an additional 1 mL of platelet rich plasma for lab analysis of platelet concentration using a standard lab automated analyzer. This extra 1 ml of whole blood will be drawn at the same time that the 35 ml described above is drawn.

The 3 ml of platelet rich plasma will be injected into the subject's Achilles tendon. The specimens will not be kept or stored. The blood will be analyzed on the same day as the procedure is being performed. This will not require storing of the specimen and prevent erroneous labeling of platelet concentration with a different subject.

After the injections, the subject will rest for 5 minutes. Participants will be given acetaminophen for "as-needed" analgesia and will be telephoned after 3 days to inquire about side effects or adverse events. Subjects will be placed in a boot for two weeks with gradual return to activity. Subjects will also be provided crutches to be non-weight bearing for 24 hours.

Data and Safety Monitoring Plan The data and safety monitoring plan to be implemented in this study consists, in part, of a monthly staff meeting to discuss subject enrollment, safety, and retention. These meetings are intended to monitor participant study flow from initial eligibility assessment to study completion. Standing agenda items for these meetings will be side effects, adverse events and participant retention.

Unanticipated adverse events and complications will be evaluated and treated if necessary by the Principal Investigator and the primary Co-Investigator.

In addition, the following processes will help ensure the timely detection, evaluation and treatment:

1. The Principal Investigator and the primary Co-Investigator will screen subjects for adverse events prior to treatment with PRP. Standardized forms will be used for monitoring and reporting of adverse events. The PI will be immediately available to staff via cell phone in case of a serious adverse event. The PI will immediately report serious adverse events to the UW Research Subjects Advocate using standardized forms. Reports will be made using the subject identification number without other identifying information.
2. Autologous injection of PRP has been found to be safe. The system being used was chosen for its closed system to prevent contamination and for its ease of use. Although safe, internal monitoring of PRP injection safety will also be performed. The study coordinator will assess each PRP injection subject 3 days after treatment with the following question during a brief telephone interview: "Do you think that you have had any side effects from the injection you've received?" [If "Yes"] "Please tell me more about that." Information regarding side effects and adverse events will be made available to the PI, who will decide if the subject requires further medical care.

Investigators do not expect serious adverse events (SAEs) but are well equipped to manage them. Investigators have not seen significant adverse events in combined (UW Radiology and Sports Medicine) clinic use of PRP. Subjects with reactions to acetaminophen or injections have the option to call study personnel at any time. The PI and the primary Co-Investigator will share on-call duty for subjects with adverse events through a pager on a 24/7 basis. Subjects who require significant evaluation and care will be referred to the UW Hospital Emergency Department.

Adverse events from a diagnostic ultrasound are extremely unlikely because ultrasound is considered to have non-significant risk by the FDA. All study procedures will be monitored and documented, and in the unlikely situation where an adverse event occurs, it will be followed to resolution.

The PI(a Board-Certified radiologist) will assess whether the findings should be reported to subjects. Findings that would be reported are those considered clinically relevant. Findings that are considered normal variants (eg. variant anatomy) or clinically insignificant (eg. simple hepatic cyst) will not be reported. Clinically relevant findings will be reported to the subject within 24 hours of the scan, and will also be reported to the subject's physician according to whether the subject has indicated a desire for this in the consent form.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years, inclusive
2. diagnosis of moderate to severe AT, confirmed by Dr. Wilson using clinical symptoms and exam findings consistent with chronic AT (>6 month duration) - which includes pain while palpating the intratendinous swelling part of the Achilles tendon and relief of pain when tendon placed under tension - and pre-procedure US
3. self-reported AT-related pain for at least 6 months and VAS (Visual Analog Scale) pain >5 (0-10 scale)
4. self-reported failure of eccentric exercise protocol (at least 75% completion)
5. self-reported failure of at least 2 of the 3 most common treatments for AT (NSAIDS, rest/ice or taping)
6. patient considered surgery but decided to wait and/or refused surgery -

Exclusion Criteria:

1. bilateral AT
2. insertional AT
3. local steroid injection within 6 weeks or physical therapy within 4 weeks
4. inability to comply with follow-up criteria
5. history of surgery on the Achilles tendon or systemic diseases (general inflammatory diseases such as rheumatologic disorders and diabetes)
6. daily use of opioids for pain
7. anticoagulation or immunosuppressive therapy
8. intent to use NSAIDs or steroids
9. self-reported pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Structure and Biomechanical function | 12 weeks
  Primary outcome measure: Estimate ultrasound based changes consistent with disease modification in two ways:
  1. conventional ultrasound to assess Achilles tendon thickness, neovascularity, and hypoechogenicity.
  2. estimate AE and SWI variability and the correlations of AE and SWI with conventional ultrasound measures to plan future research.

SECONDARY OUTCOMES:
Quality of Life Assessment | 12 weeks
  Secondary outcome measure: Quality of life will be assessed with the VISA-A validated questionnaire of pain and function of the Achilles tendon. This measure will be administered at three time points.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lee, MD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States